CLINICAL TRIAL: NCT02670330
Title: An Open Label Multi-Center Extension Study to Evaluate the Long-term Safety of Zorblisa™ (SD-101-6.0) in Patients With Epidermolysis Bullosa
Brief Title: Open Label Extension Study to Evaluate the Long-term Safety of Zorblisa (SD-101-6.0) in Patients With Epidermolysis Bullosa
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Sponsor voluntarily recalled SD-101 and terminated the study due to GMP deficiencies identified during an FDA inspection at the site of the manufacturer.
Sponsor: Scioderm, Inc. (Industry)
Collaborators: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SD-006; 2014-005679-96 (EudraCT Number)
Record Dates: First submitted 2015-07-28; First posted 2016-02-01 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Epidermolysis Bullosa
Keywords: Amicus Therapeutics; Scioderm, Inc.; Simplex; Recessive Dystrophic; Junctional non-Herlitz; Epidermolysis Bullosa; SD-101 6%; SD-101-6.0; Allantoin 6%; Zorblisa
MeSH Terms: conditions — Epidermolysis Bullosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental: SD-101-6.0 cream (Experimental): All participants (or their caregivers) applied SD-101-6.0 cream topically once a day to the entire body for a period of up to 36 months.
  Interventions: Drug: SD-101-6.0 cream

INTERVENTIONS:
Drug: SD-101-6.0 cream — SD-101 is a white, crystalline powder that is formulated within an odorless, soft, white cream base. SD-101-6.0 cream contains allantoin, a diureide glyoxylic acid, at a concentration of 6% and other excipients.
  Other Names: Zorblisa; SD-101

SUMMARY:
The study aimed to assess the long-term safety of topical use of Zorblisa (SD-101-6.0) in participants with Epidermolysis Bullosa (EB).

DETAILED DESCRIPTION:
This was an open label, multi-center extension study to assess the long-term safety of topically applied SD-101-6.0 in participants with simplex, recessive dystrophic, and junctional non-Herlitz EB. SD-101-6.0 was applied topically once a day to the entire body. The planned duration of treatment with SD-101-6.0 for Study SD-006 was up to 48 months, with a safety follow-up period of 30 days; however, the study was terminated early by the sponsor. The maximum study duration completed by at least 1 participant, treatment and safety follow-up, was 37 months.

Participants who successfully completed Study SD-005 had the option to rollover into Study SD-006. The screening/baseline visit (Visit 1) occurred at Visit 5 (approximately 90 days from baseline) of Study SD-005. The Body Surface Area (BSA) assessments of lesional skin and wound burden performed at Visit 5 (approximately 90 days from baseline) for Study SD-005 were utilized as the baseline assessments for Study SD-006. Participants returned for follow-up visits at Month 1 then every 3 months.

At each visit, assessments included BSA of lesional skin and wound burden. For target wounds that are not closed by the end of Study SD-005, the ARANZ picture and calculation of target wound area at the final visit for Study SD-005 was used as the baseline area size of the target wound for Study SD-006. These unhealed target wounds from Study SD-005 were assessed via ARANZ SilhouetteStar™ at each subsequent scheduled visit until the target wound was documented as closed. Closed wounds were assessed for scarring.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Form signed by the participant or participant's legal representative; if the participant was under the age of 18 but capable of providing assent, signed assent from the participant.
* Participant (or caretaker) must have been willing to comply with all protocol requirements.
* Participants who completed the SD-005 study (on study drug at Visit 5, approximately 90 days from baseline).

Exclusion Criteria:

* Participants who did not meet the entry criteria outlined above.
* Pregnancy or breastfeeding during the study. (A urine pregnancy test was performed at the final visit for Study SD-005 for female participants of childbearing potential and repeated at screening/baseline visit of Study SD-006 if these visits did not occur on the same day).
* Female participants of childbearing potential who were not abstinent or not practicing a medically acceptable method of contraception.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2015-06-09 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Amicus Therapeutics
Locations (30):
- United States (15):
  - Phoenix, Arizona
  - Redwood City, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Chicago, Illinois
  - Minneapolis, Minnesota
  - Columbia, Missouri
  - St Louis, Missouri
  - East Setauket, New York
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - San Antonio, Texas
  - Seattle, Washington
- Australia (2):
  - Kogarah, New South Wales
  - Parkville, Victoria
- Salzburg, Austria
- France (3):
  - Nice
  - Paris
  - Toulouse
- Germany (2):
  - Freiburg im Breisgau
  - Hanover
- Tel Aviv, Israel
- Kaunas, Lithuania
- Groningen, Netherlands
- Warsaw, Poland
- Belgrade, Serbia
- Madrid, Spain
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 152 participants with epidermolysis bullosa (EB) were enrolled between 9 June 2015 and 5 July 2017 in this open-label, multi-center extension study. All enrolled participants had previously completed Study SD-005 (NCT02384460).
Pre-assignment Details: Analysis groups were defined based on prior treatment in Study SD-005: 77 participants who received placebo were allocated to the 'Placebo to Zorblisa™ (SD-101-6.0)' group and 75 participants who received SD-101-6.0 were allocated to the 'SD-101-6.0 to SD-101-6.0' group. All participants received SD-101-6.0 upon enrolling in Study SD-006.
Groups:
- SD-101-6.0 to SD-101-6.0: Participants who received SD-101-6.0 in Study SD-005 continued to receive SD-101-6.0 in this open label extension study. SD-101-6.0 was applied topically once a day to the entire body.
- Placebo to SD-101-6.0: Participants who received placebo in Study SD-005 received SD-101-6.0 in this open-label extension study. SD-101-6.0 was applied topically once a day to the entire body.
Period: Overall Study
Arm/Group | SD-101-6.0 to SD-101-6.0 | Placebo to SD-101-6.0
Started | 75 | 77
Received At Least 1 Dose Of Study Drug (Safety Population) | 75 | 77
Completed | 0 | 0
Not Completed | 75 | 77
Not completed — Protocol Deviation | 1 | 0
Not completed — Study Terminated By Sponsor | 36 | 43
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 34 | 29
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all participants who rolled over from Study SD-005.
Groups:
- Total: Total of all reporting groups
Arm/Group | SD-101-6.0 to SD-101-6.0 | Placebo to SD-101-6.0 | Total
Number analyzed (Participants) | 75 | 77 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.18 (13.381) | 14.36 (13.599) | 14.27 (13.447)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 45 | 73
  Male | 47 | 32 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 13 | 18
  Not Hispanic or Latino | 67 | 60 | 127
  Unknown or Not Reported | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 65 | 63 | 128
  Black or African-American | 4 | 3 | 7
  Asian | 3 | 7 | 10
  American Indian or Alaskan Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific | 0 | 0 | 0
  Other | 1 | 1 | 2
  Unknown | 2 | 3 | 5
EB Type [Count of Participants; unit: Participants]
  Simplex | 9 | 7 | 16
  Recessive Dystrophic | 53 | 56 | 109
  Junctional Non-Herlitz | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as adverse events that started or worsened on or after baseline visit.
Time Frame: From baseline to 30 days after last application of study drug (up to a maximum of 37 months)
Population: Safety Population: all participants who applied/were administered the study drug at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | SD-101-6.0 to SD-101-6.0 | Placebo to SD-101-6.0
Number analyzed (Participants) | 75 | 77
Participants
  Any TEAE | 51 | 58
  Any TEAE Related To Study Drug | 8 | 17
  Any Fatal TEAE | 0 | 0
  Any Serious TEAE | 11 | 14
  Any TEAE Leading To Discontinuation | 2 | 3

2. Secondary Outcome: Change From Baseline In Body Surface Area Index (BSAI) Of Lesional Skin Up To Month 30
Description: Lesional skin was defined as areas that contained any of the following: blisters, erosions, ulcerations, scabbing, bullae, or eschars, as well as areas that were weeping, sloughing, oozing, crusted, or denuded. The percentage, ranging from 0% to 100%, of affected body surface area (BSA) was recorded for each defined body region (that is, head/neck, upper limbs, trunk [includes groin], and lower limbs), multiplied by the weighting factor, then summed for all body regions to calculate the BSAI that would range from 0% to 100%. The BSA for lesional skin was to be assessed by the same study physician on each visit for a particular participant. The mean change from baseline in BSAI was assessed every 3 months. Only participants with data available for analysis at each time point are presented.
Time Frame: Baseline, up to Month 30
Population: Intent-to-treat (ITT) population: all participants who rolled over from Study SD-005 and had data available for analysis at each specified time point.
Measure: Mean (Standard Deviation); unit: Percentage of BSAI
Arm/Group | SD-101-6.0 to SD-101-6.0 | Placebo to SD-101-6.0
Number analyzed (Participants) | 75 | 77
Percentage of BSAI
  Month 1: number analyzed (Participants) | 70 | 71
  Month 1 | -0.76 (4.185) | -0.54 (5.398)
  Month 3: number analyzed (Participants) | 69 | 66
  Month 3 | -1.87 (5.999) | -1.21 (6.457)
  Month 6: number analyzed (Participants) | 64 | 60
  Month 6 | -1.77 (6.015) | -1.35 (6.813)
  Month 9: number analyzed (Participants) | 61 | 56
  Month 9 | -2.48 (9.436) | 0.31 (10.117)
  Month 12: number analyzed (Participants) | 52 | 50
  Month 12 | -3.35 (9.566) | 0.44 (10.327)
  Month 15: number analyzed (Participants) | 35 | 29
  Month 15 | -1.90 (7.337) | 2.15 (12.546)
  Month 18: number analyzed (Participants) | 25 | 26
  Month 18 | -2.46 (5.275) | -4.24 (8.207)
  Month 21: number analyzed (Participants) | 18 | 16
  Month 21 | -3.06 (5.869) | -1.58 (10.442)
  Month 24: number analyzed (Participants) | 11 | 7
  Month 24 | -1.63 (5.647) | -0.64 (5.981)
  Month 27: number analyzed (Participants) | 6 | 6
  Month 27 | -1.87 (4.405) | -0.16 (6.514)
  Month 30: number analyzed (Participants) | 3 | 5
  Month 30 | -2.77 (5.465) | 3.37 (10.706)

3. Secondary Outcome: Change From Baseline In BSAI Of Total Body Wound Burden Up To Month 30
Description: A wound was defined as an open area on the skin (that is, epidermal covering disrupted). Total body wound burden was calculated using BSAI; the percentage, ranging from 0% to 100%, of affected BSA was recorded for each defined body region (that is, head/neck, upper limbs, trunk [includes groin], and lower limbs), multiplied by the weighting factor, then summed for all body regions to calculate the BSAI that would range from 0% to 100%. The BSAI for total body wound burden was to be assessed by the same study physician at each visit for a particular participant.
  The mean change from baseline in total body wound burden was assessed every 3 months. Only participants with data available for analysis at each time point are presented.
Time Frame: Baseline, up to Month 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of BSAI
Arm/Group | SD-101-6.0 to SD-101-6.0 | Placebo to SD-101-6.0
Number analyzed (Participants) | 75 | 77
Percentage of BSAI
  Month 1: number analyzed (Participants) | 70 | 71
  Month 1 | -1.75 (4.891) | 0.07 (4.044)
  Month 3: number analyzed (Participants) | 69 | 66
  Month 3 | -1.52 (5.343) | -0.80 (3.001)
  Month 6: number analyzed (Participants) | 64 | 60
  Month 6 | -1.54 (4.322) | -0.48 (3.595)
  Month 9: number analyzed (Participants) | 61 | 56
  Month 9 | -1.82 (6.083) | -0.42 (3.586)
  Month 12: number analyzed (Participants) | 52 | 50
  Month 12 | -1.38 (5.497) | -0.13 (3.211)
  Month 15: number analyzed (Participants) | 35 | 29
  Month 15 | -0.15 (4.511) | 0.26 (3.030)
  Month 18: number analyzed (Participants) | 25 | 26
  Month 18 | -1.12 (3.053) | -1.31 (4.665)
  Month 21: number analyzed (Participants) | 18 | 16
  Month 21 | -1.44 (3.150) | -0.28 (5.507)
  Month 24: number analyzed (Participants) | 11 | 7
  Month 24 | -0.68 (3.890) | -0.01 (2.898)
  Month 27: number analyzed (Participants) | 6 | 6
  Month 27 | -0.43 (2.924) | 0.31 (3.615)
  Month 30: number analyzed (Participants) | 3 | 5
  Month 30 | -1.55 (2.883) | 1.69 (5.933)

ADVERSE EVENTS:
Time Frame: From baseline to 30 days after last application of study drug (up to a maximum of 37 months).
Arm/Group | SD-101-6.0 to SD-101-6.0 | Placebo to SD-101-6.0
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/77
Serious Adverse Events (participants affected / at risk) | 11/75 | 14/77
Other Adverse Events (participants affected / at risk) | 44/75 | 51/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SD-101-6.0 to SD-101-6.0 (N=75) | Placebo to SD-101-6.0 (N=77)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Pericarditis (Cardiac disorders) | 1 | 0
Congenital megaureter (Congenital, familial and genetic disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 1
Gastroenteritis clostridial (Infections and infestations) | 0 | 1
Implant site infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Skin bacterial infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 2
Staphylococcal skin infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Wound infection bacterial (Infections and infestations) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 1
Stoma site extravasation (Injury, poisoning and procedural complications) | 0 | 1
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Feeding intolerance (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Intermittent explosive disorder (Psychiatric disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SD-101-6.0 to SD-101-6.0 (N=75) | Placebo to SD-101-6.0 (N=77)
Anaemia (Blood and lymphatic system disorders) | 5 | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2
Epidermolysis bullosa (Congenital, familial and genetic disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 2
Oesophageal dilatation (Gastrointestinal disorders) | 2 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 3 | 4
Toothache (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3
Pain (General disorders) | 2 | 2
Pyrexia (General disorders) | 5 | 10
Systemic inflammatory response syndrome (General disorders) | 0 | 2
Bronchitis (Infections and infestations) | 5 | 1
Cellulitis (Infections and infestations) | 3 | 0
Cystitis (Infections and infestations) | 2 | 0
Eye infection (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 0 | 3
Influenza (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 10 | 6
Otitis media (Infections and infestations) | 3 | 0
Pharyngitis streptococcal (Infections and infestations) | 2 | 4
Pyoderma (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 4 | 1
Skin bacterial infection (Infections and infestations) | 4 | 4
Skin infection (Infections and infestations) | 6 | 12
Staphylococcal skin infection (Infections and infestations) | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 5
Urinary tract infection (Infections and infestations) | 2 | 1
Viral rash (Infections and infestations) | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 2
Wound infection (Infections and infestations) | 3 | 6
Wound infection bacterial (Infections and infestations) | 2 | 5
Wound infection pseudomonas (Infections and infestations) | 2 | 2
Wound infection staphylococcal (Infections and infestations) | 2 | 3
Corneal abrasion (Injury, poisoning and procedural complications) | 2 | 2
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0
Wound (Injury, poisoning and procedural complications) | 3 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 6
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
Results are presented for all participants who received SD-101-6.0 before the early termination of the study on 4 June 2018. The maximum study duration completed by at least 1 participant was 37 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT02670330/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT02670330/SAP_001.pdf